CLINICAL TRIAL: NCT04458649
Title: Continuous Glucose Monitoring in Infants
Status: Recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Dr Jane Kim, Professor of Pediatrics, University of California, San Diego
Other Study IDs: 191263
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Neonatal Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- No increased risk of hypoglycemia: Infants born with no obvious risk factors for hypoglycemia in the neonatal period.
  Interventions: Device: Dexcom continuous glucose monitor
- Increased risk of hypoglycemia: Infants considered at increased risk for hypoglycemia after birth including the following criteria:
  * Infant born to a diabetic mother
  * Very large for gestational age (VLGA) infant with weight >97%
  Interventions: Device: Dexcom continuous glucose monitor

INTERVENTIONS:
Device: Dexcom continuous glucose monitor — Measurement of interstitial glucose

SUMMARY:
The purpose of this study is to employ continuous glucose monitoring to measure glucose profiles in newborn infants.

DETAILED DESCRIPTION:
We will place a continuous glucose monitor on the infant within 2 hours of birth and record blood glucose values every 5 minutes via the monitor; in addition, the infant will receive blood glucose checks via heel stick according to the standard hospital glucose monitoring protocol.

ELIGIBILITY:
Inclusion Criteria:

* Mother at least 18 years of age
* Infants born either appropriate for gestational age (AGA) or large for gestational age (LGA)
* Skin fold over superior gluteus area at least 1 inch in thickness as measured by skin calipers

Exclusion Criteria:

* Infants born small for gestational age (SGA)
* Infant birth weight <2.5 kg
* Infant BMI <10th percentile on Olsen chart
* Infants born <38 weeks gestation
* Infants with concern for intrauterine growth restriction (IUGR) and short femur length based on ultrasound
* Mother is non-English speaking

Ages: 1 Hour to 2 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Mother/infant dyads will be admitted at UCSD Jacobs Medical Center for antepartum and postpartum care.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Time spent with glucose <40 mg/dL | The device will be worn from about 2 hours after birth until hospital discharge, up to a maximum of 10 days. It will be removed sooner if required for medical care or if the parent requests removal.
  The Dexcom continuous glucose monitors measure interstitial fluid glucose values every 5 minutes. Data obtained from the Dexcom tracings will allow us to quantify how much time both infants with no risk for hypoglycemia (defined here as <40 mg/dL) and those with risk factors for hypoglycemia spend at a blood glucose of <40 mg/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Kim, MD, Principal Investigator — University of California San Diego/Rady Children's Hospital
Locations (1):
- UCSD Medical Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thompson-Branch A, Havranek T. Neonatal Hypoglycemia. Pediatr Rev. 2017 Apr;38(4):147-157. doi: 10.1542/pir.2016-0063. PMID 28364046
- [Background] Adamkin DH. Neonatal hypoglycemia. Curr Opin Pediatr. 2016 Apr;28(2):150-5. doi: 10.1097/MOP.0000000000000319. PMID 26780301
- [Background] Straussman S, Levitsky LL. Neonatal hypoglycemia. Curr Opin Endocrinol Diabetes Obes. 2010 Feb;17(1):20-4. doi: 10.1097/MED.0b013e328334f061. PMID 19952738